CLINICAL TRIAL: NCT05531214
Title: A Comparative Effectiveness Study to Assess the Impact of a Multidisciplinary Cardiorenal Care Team to Assist Primary Care Clinicians in Managing Patients With Heart Failure and Chronic Kidney Disease vs Usual Care.
Brief Title: Creating A Cardiorenal Multidisciplinary Team for Management HF and CKD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Gurusher Panjrath, Professor of Medicine, Fellowship Director of Nephrology, Cardiorenal Program Director, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NCR224155
Record Dates: First submitted 2022-06-10; First posted 2022-09-07 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure; Chronic Kidney Diseases
MeSH Terms: conditions — Heart Failure; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Our pragmatic randomized controlled trial will firstly identify primary care clinicians (PCCs) currently working at the George Washington University Medical Faculty Associates (GW-MFA) who care for adult patients diagnosed with both heart failure with a reduced ejection fraction (HFrEF) and chronic kidney disease (CKD). 164 patients who meet our inclusion criteria will be first identified via their respective PCCs at the GW-MFA. These PCCs will be randomized to the control and intervention arms, and the intervention arm will be receiving recommendations from a multidisciplinary team of cardiologists and nephrologists.
Who Masked: Participant
Masking Description: These primary care clinicians will then be block randomized using a 1:1 ratio to either arm of treatment utilizing random number generation. Primary care clinicians will be stratified by the size of their individual practices, and patients will be stratified by EF prior to their enrollment to balance the representation of patients with HFrEF (EF < 50%) and heart failure with mildly reduced ejection fraction (HFmrEF) (EF 41-49%), respectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients randomized based on their primary care clinician to a co-localized care with a telemedicine-based cardiorenal multidisciplinary team (cardiologist, nephrologist, and research coordinators) providing guidance and recommendations to the primary care clinician.
  Interventions: Behavioral: Multidisciplinary Care Coordination Team
- Control (No Intervention): Patients randomized to the control group will proceed with usual care with a primary care clinician making referrals to a cardiologist or nephrologist "for-cause" as determined by the primary care clinician, to ultimately assess the rates of improvement in the implementation of GDMT.

INTERVENTIONS:
Behavioral: Multidisciplinary Care Coordination Team — The intervention group will be patients whose primary care clinicians will be receiving guidance and recommendations from the multidisciplinary team consisting of cardiologists, nephrologists, and specialty pharmacists.
  Arms: Intervention

SUMMARY:
Several drugs have been labeled as guideline-directed-medical therapies (GDMT) to improve overall health outcomes and slow the progression of disease in patients with heart failure (HF). Although scientific trials have deemed these drugs to be successful, many HF patients have been unable to either get started on the appropriate drug regimens or be optimized on the doses required to show substantial benefit, particularly in those who also suffer from chronic kidney disease (CKD). This is largely due to the current health care delivery model that requires a primary care clinician or general internist to refer patients to heart failure specialists and nephrologists. The specialty care itself then requires even more coordination resulting in patients getting lost to follow-up, physicians losing track of recommendations from different clinics, and too many separate electronic medical documentations to consolidate prior to deciding on what medication is appropriate at one thirty-minute outpatient visit. This study plans to create a new, virtual cardio-renal multidisciplinary team including a heart failure specialist and nephrologist to ease the coordination of care and consequently show a better implementation of GDMT in patients with HF and CKD when comparing those rates to the traditional referral-based way that these medications get prescribed.

DETAILED DESCRIPTION:
Major advancements have occurred in guideline-directed medical therapies (GDMT) for heart failure (HF) over the last decade. Various classes of drugs including beta-adrenergic receptor blockers, renin-angiotensin system inhibitors, sodium-glucose co-transporter inhibitors, etc. have demonstrated significant improvement in the quality of life, prevention of recurrent hospitalizations for HF, and reduction in overall morbidity and mortality. However, despite the billions of healthcare dollars and additional clinical resources invested into developing these evidence-based treatment regimens, a substantial proportion of the affected patient populations remains undertreated worldwide rendering GDMT unrealistic to implement broadly, particularly in the subgroup of patients with concomitant chronic kidney disease (CKD).

Several deterrents contribute to the low implementation rates of GDMT in HF with CKD including clinicians' therapeutic inertia and fear of inducing harm, poor coordination of care between inpatient and outpatient titration of medications, fragmented healthcare models, inaccessibility to specialists' support, and high-cost burden deeming certain medications unaffordable. These factors also primarily affect minority communities, patients among the lower socioeconomic strata, and individuals with limited health literacy who are unequally affected by higher rates of HF with CKD. Although current research can both qualify and quantify the benefits of the medications, minimal treatment prototypes exist to ensure that patients have and maintain access to these therapies, the frequent follow-up visits, and the surveillance screenings required to monitor long-term symptoms and potential medication side-effects.

This study aims to compare the effects of a co-localized multidisciplinary cardiorenal team supporting a primary care clinician versus the traditional referral-based care model, on the implementation rates of GDMT in patients with specifically heart failure with reduced ejection fraction (HFrEF) and CKD. Investigators will conduct a single-center pragmatic randomized controlled trial that will compare the following approaches:

1. Co-localized care with a telemedicine-based cardiorenal multidisciplinary team (cardiologist, nephrologist, and research coordinators) providing guidance and recommendations to the primary care clinician 2. A control group of usual care with a primary care clinician making referrals to a cardiologist or nephrologist "for-cause" as determined by the primary care clinician, to ultimately assess the rates of improvement in the implementation of GDMT. The research coordinators will also play a crucial role in identifying financial barriers, circumventing insurance and prior authorization issues, as well as monitoring medication side-effect profiles and potential drug-to-drug interactions as they pertain to each individual patient involved in the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* History of HF with reduced ejection fraction (HFrEF) or ejection fraction (EF) <50% and chronic kidney disease (CKD) with estimated glomerular filtration rate (eGFR) < 60cc/min/1.73m2

Exclusion Criteria:

* Patients < 18 years of age
* Patients with a heart or kidney transplant
* Patients on dialysis at the time of enrollment
* Pregnant
* Non-English speaking
* Patients that are unable to understand the process of the study and consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Difference in rate of sodium glucose co-transporter 2 inhibitors (SGLT2i) | 6 months
  Given that increased SGLT2i is likely to be the major driver of improved clinical outcomes in patients with heart failure and chronic kidney disease, the primary outcome of interest is the difference in rate of SGLT2i use between multidisciplinary care model versus usual care model at 3 months and 6 months.

SECONDARY OUTCOMES:
Quality of life of patients-Kidney Disease Questionnaire | 6 months
  Quality of life will be measured by a score at baseline, 3-months, and 6-months, using the Kidney Disease and Quality of Life survey (KDQOL-36).
Quality of life of patients-Cardiomyopathy Questionnaire | 6 months
  Quality of life will be measured by a score at baseline, 3-months, and 6-months, using the Cardiomyopathy Questionnaire (Kansas City) (KCCQ-12).
Heart failure hospitalizations | 6 months
  Heart failure hospitalizations, ≥40% sustained decline in kidney function, need for maintenance dialysis or a kidney transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Janai Rangaswami, MD, Principal Investigator — Fellowship program director for the Division of Nephrology, Director of the cardiorenal program
Locations (1):
- George Washington University Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No